CLINICAL TRIAL: NCT04096534
Title: Normotonic Partial Nephrectomy as Novel Approach in Treating Small Renal Masses
Acronym: NORPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Vladislav Osetnik, Principal Investigator, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NORPN
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Renal Malignant Tumor; Renal Tumor
Keywords: partial nephrectomy; zero ischaemia; renal function
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normotonic partial nephrectomy (Experimental): Performing a partial nephrectomy under normal body blood pressure
  Interventions: Procedure: Normotonic partial nephrectomy
- Hypotonic partial nephrectomy (Active Comparator): Performing a partial nephrectomy under hypotonic body blood pressure
  Interventions: Procedure: Hypotonic partial nephrectomy

INTERVENTIONS:
Procedure: Normotonic partial nephrectomy — partial nephrectomy performing with avoidance of hypotension: mean blood pressure more or equal 65 mm Hg
  Arms: Normotonic partial nephrectomy
Procedure: Hypotonic partial nephrectomy — partial nephrectomy performing with using of medical hypotension; avoidance of hypertension: mean blood pressure less than 65 mmHg
  Arms: Hypotonic partial nephrectomy

SUMMARY:
This study evaluates novel surgical approach in treating small renal masses. Half of participants will undergo hypotonic zero-ischaemia partial nephrectomy (standard of care), while the other half will undergo normotonic zero-ischaemia partial nephrectomy (experimental method).

DETAILED DESCRIPTION:
Partial nephrectomy is believed to be the gold standard for treating small renal masses (SRM). The warm ischaemia and hypotonic zero-ischaemia approach are widely used techniques of care. But they have some negative effects according to renal function (RF) after surgery. We decided to compare influence of arterial blood pressure (normotension or hypotension) during partial nephrectomy on RF.

A single-center prospective study comparing normotonic and hypotonic partial nephrectomy will be conducted.

The design involves random allocation of eligible patients to normotonic or hypotonic partial nephrectomy group in 1:1 ratio.

Experimental group - normotonic partial nephrectomy (avoidance of hypotension: mean blood pressure more or equal 65 mm Hg).

Control group - hypotonic partial nephrectomy (using medical hypotension; avoidance of hypertension: mean blood pressure less than 65 mmHg

According to preliminary calculations, taking into account type I error of 5% and power of 80%, 100 patients should be included in the study. In order to compensate for data loss, the estimated sample size is increased by 10%. As a result, the total sample size is 100 +10 = 110 patients (55 patients for each group). The expected duration of the study is 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Suspected by computed tomography or another instrumental method renal mass
* Clinical stage T1-2N0-2M0-1 (distant metastases must be resectable)
* Indications for partial nephrectomy
* Eastern Cooperative Oncology Group status 0-2
* At least 18 years of age
* Written informed consent

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or comply with the study protocol
* Pregnancy or breast feeding
* Medical contraindications for surgical treatment
* Synchronous or metachronous malignancy
* Non-resectable distant metastases
* The patient's refusal to perform research procedures.
* Refusal of the patient to continue participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-05-07 (Actual)

PRIMARY OUTCOMES:
Renal function | within the first 3 month after surgery
  glomerular filtration rate calculation (mL/min), nephroscintigraphy
Blood loss | enrollment
  Volume of intraoperative blood loss (ml)

SECONDARY OUTCOMES:
Disease-free survival | 1 year after last patient enrolled
  Survival without local or systemic recurrence (months)
Resection margins status | enrollment
  Evaluating of resection margins status (positive/negative)

CONTACTS AND LOCATIONS:
Overall Officials: Imran Dzhalilov, MD, Study Director — Saint Petersburg State University, Russia; Vladislav Osetnik, MD, Principal Investigator — Saint Petersburg State University, Russia; Batyrbek Aslanov, PhD, Study Chair — Mechnikov North-West State Medical University
Locations (1):
- State University Clinic, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No
We are not planning to share personal patient data